CLINICAL TRIAL: NCT05468450
Title: Three-year Outcomes of a RCT Comparing EVLA Versus Polidocanol Foam in the Treatment of SSV Insufficiency (FOVELASS Study, by the French Society of Phlebology)
Brief Title: RCT Comparing EVLA Versus Polidocanol Foam in the Treatment of SSV Insufficiency
Acronym: FOVELASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Societe Francaise de Phlebologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01943-44
Record Dates: First submitted 2022-07-13; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Varicose Veins of Lower Limb
Keywords: small saphenous veins; varicose veins; ultrasound guided foam sclerotherapy; endovenous laser ablation
MeSH Terms: conditions — Varicose Veins | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: multicentre-RCT (11 centres) comparing ultrasound-guided-foam sclerotherapy (UGFS) and Endovenous Laser Ablation (EVLA) for treating small saphenous veins (SSV) insufficiency
Masking Description: Blinding of participants and investigators is not possible because of the obvious differences between the two treatments (a single mid-calf injection versus multiple injections for tumescent anaesthesia/laser precautions etc…).
  A blind third-party check was carried out, only at 3 years, and those assessors were completely independent of the study and blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided-foam sclerotherapy (UGFS) (Active Comparator): Injection of Polidocanol foam into SSV
  Interventions: Drug: Ultrasound-guided-foam sclerotherapy (UGFS) using Polidocanol sclerosant
- Endovenous Laser Ablation (EVLA) (Active Comparator): Ablation of SSV using laser energy
  Interventions: Device: Endovenous Laser Ablation (EVLA)

INTERVENTIONS:
Drug: Ultrasound-guided-foam sclerotherapy (UGFS) using Polidocanol sclerosant — Direct injection Foam sclerotherapy
  Other Names: Foam sclerotherapy
  Arms: Ultrasound-guided-foam sclerotherapy (UGFS)
Device: Endovenous Laser Ablation (EVLA) — EVLA using a 1470nm generator and 600-micron radial fibres (Biolitec® Biomedical Technology, Jena, Germany), under tumescent local anaesthesia (TLA)
  Other Names: Laser therapy
  Arms: Endovenous Laser Ablation (EVLA)

SUMMARY:
FOVELASS is a multicentre-RCT (11 centres) comparing ultrasound-guided-foam sclerotherapy (UGFS) and Endovenous Laser Ablation (EVLA) for treating SSV insufficiency, conducted by the French Society of Phlebology.

DETAILED DESCRIPTION:
Saphenous vein insufficiency is a common finding in varicose veins cases. International guidelines currently recommend endovenous thermal ablation using laser (EVLA) or radiofrequency as first line treatment for truncal Great Saphenous Vein (GSV) incompetence in preference to Ultrasound Guided Foam Sclerotherapy (UGFS) (1,2). This GSV-based recommendation has tended to be used for treating Small Saphenous Vein (SSV) incompetence.

To date, no RCTs have directly compared UGFS and EVLA for SSV treatment. The French Society of Phlebology (SFP) decided to compare these two most utilised endovenous treatments in France in a controlled study called the FOam VErsus LAser in the SSv (FOVELASS) study, involving 13 investigators in 11 vascular medical centres.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic varicose veins (CEAP C2s-C6)
* underlying isolated SSV incompetence (SSV reflux time>0.5sec on duplex ultrasound (DUS))
* reflux involving at least 15 cm of proximal SSV
* minimal SSV diameter of 4 mm at mid-calf (luminal diameter in standing position)

Exclusion Criteria:

* SSV treatment in the preceding 3 months
* post-thrombotic disease
* deep or superficial vein thrombosis of less than 3 months duration
* coexistent ipsilateral GSV insufficiency
* morbid obesity (BMI>40)
* presence of significant arterial disease (ABPI<0.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Absence of reflux in the treated SSV segment | 3Assessed at years
  closed veins or patent veins with no reflux (>0.5sec)

SECONDARY OUTCOMES:
Treatment time | Assessed on day of treatment
  Time (in minutes) spent in undertaking each treatment
Procedure related complications | Assessed through study completion, an average of 3 years
  Any related complications arising from the procedure
Periprocedural pain score | up to four weeks
  assessed on a visual analogue score (zero = no pain, 100 = maximum pain)
Presence of visible varices | Through study completion, average of 3 years
  Reported recurrence of varicose veins
Venous symptoms questionnaire | Through study completion, average of 3 years
  Validated questionnaire scores
Revised Venous Clinical Severity Score -rVCSS | Through study completion, average of 3 years
  Validated questionnaire scores
Quality of Life questionnaire (CIVIQ) | Through study completion, average of 3 years
  Validated questionnaire scores

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Hamel-Desnos, Study Director — Institut des Varices- GHPJS Groupe Hospitalier; Matthieu Josnin, Principal Investigator — Société Française de Phlébologie

IPD SHARING:
Plan to Share IPD: No
Randomised is provided by the independent statistics centre (Cenbiotech; Dijon-France), who also analysed IPD. Investigators cannot access other centres' data.

REFERENCES:
- [Background] 9) Hamel-Desnos C., Josnin M., Allaert F.-A. Etude contrôlée randomisée de l'efficacité du laser endoveineux (1470 nm) versus échosclérothérapie à la mousse dans le traitement de l'insuffisance de la petite veine saphène. Phlébologie 2019 (72): 8-18
- [Derived] Hamel-Desnos C, Nyamekye I, Chauzat B, Gracia S, Josnin M, Abbadie F. FOVELASS: A Randomised Trial of Endovenous Laser Ablation Versus Polidocanol Foam for Small Saphenous Vein Incompetence. Eur J Vasc Endovasc Surg. 2023 Mar;65(3):415-423. doi: 10.1016/j.ejvs.2022.11.021. Epub 2022 Dec 5. PMID 36470312